CLINICAL TRIAL: NCT06443281
Title: Pain Phenotyping in Patients With Neuropathic Pain After Spinal Cord Injury
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-00134
Record Dates: First submitted 2024-04-25; First posted 2024-06-05 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injuries; Pain, Neuropathic; Nociceptive Pain; Neuropathy
MeSH Terms: conditions — Spinal Cord Injuries; Neuralgia; Nociceptive Pain | interventions — Postsynaptic Potential Summation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients with spinal cord injury with neuropathic pain
  Interventions: Diagnostic Test: Neurophysiology; Diagnostic Test: Cardiovascular test; Diagnostic Test: Experimental pain paradigms; Diagnostic Test: Quantitative sensory testing; Diagnostic Test: Clinical pain phenotype
- Patients with spinal cord injury but without neuropathic pain
  Interventions: Diagnostic Test: Neurophysiology; Diagnostic Test: Cardiovascular test; Diagnostic Test: Experimental pain paradigms; Diagnostic Test: Quantitative sensory testing
- Patients with peripheral neuropathy
  Interventions: Diagnostic Test: Neurophysiology; Diagnostic Test: Cardiovascular test; Diagnostic Test: Experimental pain paradigms; Diagnostic Test: Quantitative sensory testing; Diagnostic Test: Clinical pain phenotype
- Healthy subjects
  Interventions: Diagnostic Test: Neurophysiology; Diagnostic Test: Cardiovascular test; Diagnostic Test: Experimental pain paradigms; Diagnostic Test: Quantitative sensory testing

INTERVENTIONS:
Diagnostic Test: Neurophysiology — Pain-related evoked potentials and nerve conduction studies
Diagnostic Test: Cardiovascular test — Blood pressure control, orthostatic intolerance test, baro-reflex sensitivity, heart-rate variability
Diagnostic Test: Experimental pain paradigms — Temporal summation of pain, conditioned pain modulation
Diagnostic Test: Quantitative sensory testing — Thermal and mechanical sensory testing
Diagnostic Test: Clinical pain phenotype — Pain drawings, plus and minus signs of pain
  Groups: Patients with peripheral neuropathy; Patients with spinal cord injury with neuropathic pain

SUMMARY:
The development of neuropathic pain is one of the most debilitating sequels after a spinal cord injury (SCI). The overall aim of this study is to investigate potential underlying pathophysiological mechanisms of neuropathic pain after SCI. The functionality of the nociceptive pathway in humans as well as its plastic changes following SCI will be inferred with sophisticated sensory and pain phenotyping using quantitative sensory testing (i.e., psychophysical measures), objective neurophysiological measures of pain processing and the recording of pain-related autonomic responses (i.e., galvanic skin response, cardiovascular measures and pupil dilation). In addition, the interplay between the somatosensory and autonomic nervous system and its association with the development and maintenance of neuropathic pain after SCI will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Spinal injury cohort - general inclusion criteria:
* Aged between 18-80 years
* Traumatic and non-traumatic etiology
* Para- and tetraplegic SCI
* Complete and incomplete SCI
* SCI with and without neuropathic pain
* Additional inclusion criteria for longitudinal study:
* SCI since less than one month
* Additional inclusion criteria for cross-sectional study:
* SCI since more than one year
* Control cohorts with peripheral neuropathy:
* General inclusion criteria:
* Aged between 18-80 years
* Neurological disorder affecting the peripheral nervous system (i.e., peripheral neuropathy)
* Peripheral neuropathy with or without neuropathic pain
* Additional inclusion criteria for longitudinal study:
* Peripheral neuropathy since less than one month
* Additional inclusion criteria for cross-sectional study:
* Peripheral neuropathy since more than one year
* Control cohorts without neuropathy / healthy volunteers
* General inclusion criteria:
* Aged between 18-80 years
* No medical condition affecting the peripheral and/or central nervous system (e.g., pain, systemic disease, psychological disorder)

Exclusion Criteria:

* Inability to follow study instructions
* Pregnancy
* Medically manifested psychological disorder
* Medical condition affecting the peripheral and/or central nervous system other than the desired experimental condition (e.g., additional peripheral neuropathy in the SCI cohort)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In- and outpatients of Balgrist University Hospital Zurich
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2030-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Spinal cord injury patients: clinical pain phenotype including the spatial pain extent and pain intensity | Longitudinal: change from 1 month up to 12 months
  Pain drawings, plus and minus signs of pain
Spinal cord injury patients: clinical pain phenotype including the spatial pain extent and pain intensity | Cross-sectional: once in a chronic stage (1 year post-injury)
  Pain drawings, plus and minus signs of pain
Patients with peripheral neuropathy: clinical pain phenotype including the spatial pain extent and pain intensity | Cross-sectional: once in a chronic stage (1 year post-injury)
  Pain drawings, plus and minus signs of pain

SECONDARY OUTCOMES:
Spinal cord injury patients / healthy controls: somato-sensory evoked potentials | Longitudinal: change from 1 month up to 12 months
  Amplitude in uV
Spinal cord injury patients / healthy controls: somato-sensory evoked potentials | Longitudinal: change from 1 month up to 12 months
  Latency in ms
Spinal cord injury patients / healthy controls: contact-heat evoked potentials | Longitudinal: change from 1 month up to 12 months
  Amplitude in uV
Spinal cord injury patients / healthy controls: contact-heat evoked potentials | Longitudinal: change from 1 month up to 12 months
  Latency in ms
Spinal cord injury patients / healthy controls: N13 spinal potential | Longitudinal: change from 1 month up to 12 months
  Amplitude in uV
Spinal cord injury patients / healthy controls: N13 spinal potential | Longitudinal: change from 1 month up to 12 months
  Latency in ms
Spinal cord injury patients / healthy controls: motor neurographies | Longitudinal: change from 1 month up to 12 months
  Amplitude in mV
Spinal cord injury patients / healthy controls: motor neurographies | Longitudinal: change from 1 month up to 12 months
  Latency in ms
Spinal cord injury patients / healthy controls: motor neurographies | Longitudinal: change from 1 month up to 12 months
  Nerve conduction velocity in m/s
Spinal cord injury patients / healthy controls: sensory neurography | Longitudinal: change from 1 month up to 12 months
  Amplitude in mV
Spinal cord injury patients / healthy controls: sensory neurography | Longitudinal: change from 1 month up to 12 months
  Latency in ms
Spinal cord injury patients / healthy controls: sensory neurography | Longitudinal: change from 1 month up to 12 months
  Nerve conduction velocity in m/s
Spinal cord injury patients / healthy controls: resting blood pressure | Cross-sectional: once in a chronic stage (1 year post-injury)
  Systolic, diastolic and mean arterial pressure all in mmHg variability
Patients with peripheral neuropathy / healthy controls: changes in blood pressure after a cold pressure test | Cross-sectional: once in a chronic stage (1 year post-injury)
  Delta mmHg
Patients with peripheral neuropathy / healthy controls: changes in blood pressure after a Valsalva maneuvre | Cross-sectional: once in a chronic stage (1 year post-injury)
  Delta mmHg
Patients with peripheral neuropathy / healthy controls: changes in blood pressure after a sit-up test | Cross-sectional: once in a chronic stage (1 year post-injury)
  Delta mmHg
Patients with peripheral neuropathy / healthy controls: baro-reflex sensitivity | Cross-sectional: once in a chronic stage (1 year post-injury)
  ms/mmHg
Patients with peripheral neuropathy / healthy controls: heart rate variability | Cross-sectional: once in a chronic stage (1 year post-injury)
  RMSSD (root mean square of successive differences), high frequency/low frequency ratio
Spinal cord injury patients / healthy controls: temporal summation of pain after repetitive application of 12 pinprick stimuli | Longitudinal: change from 1 month up to 12 months
  Change in numeric rating scale of pain from the first three to the last three pinprick stimuli
Spinal cord injury patients / healthy controls: conditioned pain modulation | Longitudinal: change from 1 month up to 12 months
  Changes in pressure pain threshold (measured by an algometer in delta kg) before and during a cold water bath
Patients with peripheral neuropathy / healthy controls: temporal summation of pain after repetitive application of 12 pinprick stimuli | Longitudinal: change from 1 month up to 12 months
  Change in numeric rating scale of pain from the first three to the last three pinprick stimuli
Patients with peripheral neuropathy / healthy controls: conditioned pain modulation | Longitudinal: change from 1 month up to 12 months
  Changes in pressure pain threshold (measured by an algometer in delta kg) before and during a cold water bath
Spinal cord injury patients / healthy controls: thermal sensory testing tested with a thermode | Longitudinal: change from 1 month up to 12 months
  Warm detection threshold (°C), cold detection threshold (°C), heat pain threshold (°C), cold pain threshold (°C)
Spinal cord injury patients / healthy controls: mechanical sensory testing tested with von Frey monofilaments/pinpricks | Longitudinal: change from 1 month up to 12 months
  Mechanical detection threshold (mN)
Spinal cord injury patients / healthy controls: mechanical sensory testing tested with von Frey monofilaments/pinpricks | Longitudinal: change from 1 month up to 12 months
  Mechanical pain threshold (mN)
Spinal cord injury patients / healthy controls: mechanical sensory testing tested with von Frey monofilaments/pinpricks | Longitudinal: change from 1 month up to 12 months
  Mechanical pain sensitivity (numeric rating scale of pain 0-10)
Spinal cord injury patients / healthy controls: mechanical sensory testing tested with von Frey monofilaments/pinpricks | Longitudinal: change from 1 month up to 12 months
  Vibration detection threshold (a.u.) tested with Rydel Seiffer tuning fork
Patients with peripheral neuropathy / healthy controls: thermal sensory testing tested with a thermode | Longitudinal: change from 1 month up to 12 months
  Warm detection threshold (°C), cold detection threshold (°C), heat pain threshold (°C), cold pain threshold (°C)
Patients with peripheral neuropathy / healthy controls: mechanical sensory testing tested with von Frey monofilaments/pinpricks | Longitudinal: change from 1 month up to 12 months
  Mechanical detection threshold (mN)
Patients with peripheral neuropathy / healthy controls: mechanical sensory testing tested with von Frey monofilaments/pinpricks | Longitudinal: change from 1 month up to 12 months
  Mechanical pain threshold (mN)
Patients with peripheral neuropathy / healthy controls: mechanical sensory testing tested with von Frey monofilaments/pinpricks | Longitudinal: change from 1 month up to 12 months
  Mechanical pain sensitivity (numeric rating scale of pain 0-10)
Patients with peripheral neuropathy / healthy controls: mechanical sensory testing tested with von Frey monofilaments/pinpricks | Longitudinal: change from 1 month up to 12 months
  Vibration detection threshold (a.u.) tested with Rydel Seiffer tuning fork

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Freund, Prof. Dr. Dr., Principal Investigator — University of Zurich
Locations (1):
- Balgrist University Hospital, Zurich, Canton of Zurich, Switzerland